CLINICAL TRIAL: NCT05180305
Title: A Study to Assess Mitomic Prostate Test for Prostate Cancer Screening
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: TSH Biopharm Corporation Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: TSHMPT2001-P
Record Dates: First submitted 2021-12-12; First posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The subject will be draw for 17 ml of blood in the screening phase.The blood sample will be sent to the central laboratory for analysis by Mitomic Mitomic Prostate Test Prostate TestProstate Test to detect the 3.4 kb mitochondrial DNA deletion.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Diagnostic Test: Mitomic Prostate Test — Mitomic Prostate Test

SUMMARY:
To evaluate the diagnostic accuracy of the Mitomic Prostate Test (MPT) comparing to prostate biopsy within the intended use population.

DETAILED DESCRIPTION:
To determine the clinical performance of a blood-based test for clinically significant (CS) prostate cancer (PCa) (grade group ≥ 2) intended for use in men with prostate serum antigen levels in the 'grey zone' (PSA < 10 ng/ml). The test quantifies a previously described 3.4 kb mitochondrial DNA (mtDNA) deletion.

ELIGIBILITY:
Inclusion Criteria:

* Men of screening age (≧45) who are scheduled for prostate needle biopsy due to suspicion of prostate cancer and have a total PSA < 10ng/ml within the previous 3 months.
* Extended Sextant biopsy pattern that must include a minimum of 12 cores. MRI targeted biopsy preferred where available.
* Age, total PSA, biopsy pathology, prostate medication history, and ethnicity data must be available;
* The index biopsy must occur following and within 16 weeks of blood draw.

Exclusion Criteria:

* Subject does not undergo their prostate biopsy within 16 weeks of collection of pre-biopsy blood sample;
* Previous diagnosis of prostate cancer;
* Prostate biopsy within the previous 3 months;
* Men with a total PSA>10ng/ml within the previous 3 months;
* Provides less than the required amount of blood;
* Considered incompetent to provide informed consent;
* Does not understand and read language of informed consent;
* Age, total PSA, biopsy pathology information, medication history or ethnicity data unavailable;
* Males who are not of screening age (<45);
* Subjects whose classification as cancer positive or negative is undetermined following biopsy due to suspicious results such as Atypical Suspicious Acinar Proliferation (ASAP);
* Blood collected after index biopsy.
* Subject is taking antibiotics at the time of blood collection or has taken antibiotics within the 2 weeks prior to blood collection.

Min Age: 45 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: To investigate the mitochondrial DNA biomarker in a large group of patients suspicious for prostate cancer to evaluate the Mitomic Prostate Test (MPT)'s accuracy in target population.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Mitomic Prostate Test (MPT) | 16 weeks
  To evaluate the diagnostic accuracy of the Mitomic Prostate Test (MPT) within the intended use population.

SECONDARY OUTCOMES:
MPT compared to the current standard of care (SOC). | 16 weeks
  To evaluate optimal disease screening strategies incorporating MPT compared to the current standard of care (SOC).

CONTACTS AND LOCATIONS:
Locations (1):
- Linkou Chang Gung Memorial Hospital, Taoyuan District, Taiwan